CLINICAL TRIAL: NCT00309751
Title: Study of Pitavastatin Vs. Atorvastatin (Following Up-Titration) in Patients With Type II Diabetes Mellitus and Combined Dyslipidemia
Brief Title: Study Comparing Pitavastatin and Atorvastatin in Patients With Type II Diabetes Mellitus and Combined Dyslipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kowa Research Europe (Industry)
Responsible Party: Dragos Budinski, MD, Kowa Research Europe
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NK-104-305
Record Dates: First submitted 2005-12-08; First posted 2006-04-03 (Estimated); Results first posted 2010-01-18 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2010-02

CONDITIONS: Type II Diabetes Mellitus; Dyslipidemia
Keywords: Kowa; Type II Diabetes Mellitus; Combined Dyslipidemia; pitavastatin; NK-104; Atorvastatin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias | interventions — pitavastatin; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pitavastatin 4 mg QD (Experimental): Pitavastatin 4 mg once daily
  Interventions: Drug: Pitavastatin
- Atorvastatin 20 mg QD (Active Comparator): Atorvastatin 20 mg once daily
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Pitavastatin — Pitavastatin 4 mg QD
  Arms: Pitavastatin 4 mg QD
Drug: Atorvastatin — Atorvastatin 20 mg
  Other Names: Lipitor
  Arms: Atorvastatin 20 mg QD

SUMMARY:
The purpose of this study is to compare the efficacy and safety of pitavastatin with that of atorvastatin in patients with type II diabetes mellitus (type II DM) and combined dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Males and females (ages 18-75 years)
* Type II DM treated with oral anti-diabetic medication (sulfonylurea, metformin, glitazones, or combination therapy)
* Must have been following a restrictive diet
* Diagnosis of combined dyslipidemia

Exclusion Criteria:

* Homozygous familial hypercholesterolemia
* Conditions which may cause secondary dyslipidemia
* Uncontrolled diabetes mellitus
* Abnormal pancreatic, liver, or renal function
* Abnormal serum creatine kinase (CK) above the pre-specified level
* Significant heart disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2005-12; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dragos Budinski, Med Dr., Study Director — Kowa Research Europe
Locations (35):
- Denmark (3):
  - CCBR Aalborg, Aalborg
  - CCBR A/S, Ballerup Municipality
  - CCBR Vejle, Vejle
- Germany (5):
  - Gemeinschaftspraxis am Bahnhof, Berlin-Spandau
  - Pharmakologisches Studienzentum Chemnitz, Chemnitz
  - Internistische Diabetische Schwerpunktpraxis Dr., Frankfurt am Main
  - Internistische Gemeinschaftspraxis, Mainz
  - Gemeinschaftspraxis Dr. Senftleber, Dr. Kohler, Messkirch
- India (5):
  - Bhagwan Mahaveer Jain Heart Centre, Bangalore
  - Sri Ramachandra Medical College Hospital, Chennai
  - Apollo Hospitals, Hyderabaad
  - CARE Group of Hospitals, Hyderabaad
  - PD Hinduja Hospital, Mumbai
- Netherlands (8):
  - Andromed Breda, Breda
  - Andromed Eindhoven, Eindhoven
  - Andromed Noord, Groningen
  - Andromed Leiden, Leiden
  - Andromed Nijmegen, Nijmegen
  - Andromed Rotterdam, Rotterdam
  - Andromed Oost, Velp
  - Andromed Zoetermeer, Zoetermeer
- Poland (10):
  - Podlaski Osrodek Kardiologii, Bialystok
  - NZOZ GCP Dobra Praktyka Lekaska, Gruziadz
  - NZOZ Terapia Optima, Katowice
  - NZOZ Centrum, Poradnia Kardiologiczna, Siedlce
  - Spec. Gab. Lek. Internistyczno-Kardiologicznly, Tarnów
  - Woj.Szp.Spec.Nr 1 im. Prof. J. Gasinskiego, Tychy
  - Instytut Zywnosci i Zywienia, Warsaw
  - Lecznica PROSEN SMO, Warsaw
  - Szpital Wolski,im. Dr A. Gostynskiej, Warsaw
  - NZOZ Esculap, Przychodnia Lekary Rodzinnych, Łosice
- United Kingdom (4):
  - Synexus Reading Clinical Research Centre, Berkshire
  - Synexus Lancashire Clinical Research Centre, Lancashire
  - Synexus Merseyside Clinical Research Centre, Liverpool
  - Synexus Manchester Clinical Research Centre, Manchester

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pitavastatin 4 mg QD | Atorvastatin 20 mg QD
Started | 279 | 139
Safety Population | 275 (Subjects who received at least 1 dose of study drug) | 137 (Subjects who received at least 1 dose of study drug)
Completed | 248 | 124
Not Completed | 31 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pitavastatin 4 mg QD | Atorvastatin 20 mg QD | Total
Number analyzed (Participants) | 275 | 137 | 412
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 191 | 93 | 284
  >=65 years | 84 | 44 | 128
Age Continuous [Mean (Standard Deviation); unit: years] | 59.1 (9.21) | 59.8 (9.06) | 59.4 (9.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 59 | 179
  Male | 155 | 78 | 233

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline Low Density Lipoprotein Cholesterol (LDL-C)
Description: Percent change from baseline to Week 12 low density lipoprotein cholesterol (LDL-C)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pitavastatin 4 mg QD | Atorvastatin 20 mg QD
Number analyzed (Participants) | 274 | 136
percent change | -40.78 (19.599) | -43.25 (16.378)

2. Secondary Outcome: Number of Patients Attaining National Cholesterol Education Program (NCEP) LDL-C Target
Description: Number of patients attaining National Cholesterol Education Program (NCEP)LDL-C target (LDL-C less than 160 mg/dL) at 12 weeks
Time Frame: 12 weeks
Measure: Number; unit: Participants
Arm/Group | Pitavastatin 4 mg QD | Atorvastatin 20 mg QD
Number analyzed (Participants) | 274 | 136
Participants | 212 | 111

ADVERSE EVENTS:
Arm/Group | Pitavastatin 4 mg QD | Atorvastatin 20 mg QD
Serious Adverse Events (participants affected / at risk) | 4 | 4
Other Adverse Events (participants affected / at risk) | 29 | 22
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Pitavastatin 4 mg QD | Atorvastatin 20 mg QD
Myocardial infarction (Cardiac disorders) | 1/275 | 0/137
Tachycardia paroxysmal (Cardiac disorders) | 1/275 | 0/137
Non-cardiac chest pain (General disorders) | 0/275 | 1/137
Gastroenteritis (Infections and infestations) | 1/275 | 0/137
Alcohol poisoning (Injury, poisoning and procedural complications) | 0/275 | 1/137
Humerus fracture (Injury, poisoning and procedural complications) | 0/275 | 1/137
Blood creatinine increased (Investigations) | 1/275 | 0/137
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0/275 | 1/137
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Pitavastatin 4 mg QD | Atorvastatin 20 mg QD
Diarrhea (Gastrointestinal disorders) | 6/275 | 9/137
Nasopharyngitis (Infections and infestations) | 12/275 | 9/137
Myalgia (Musculoskeletal and connective tissue disorders) | 11/275 | 0/137
Hypertension (Vascular disorders) | 0/275 | 4/137

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days